CLINICAL TRIAL: NCT04900272
Title: Intelligent Personal Assistant for Managing Depression in Homebound Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other)
Responsible Party: Principal Investigator, Katherine O'Brien, Assistant Professor of Medicine, Division of Internal Medicine and Geriatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00212384
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Aging; Physical Dependence
Keywords: Social Isolation; Loneliness; Older Adults; Homebound
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIPA device and companion booklet (Experimental): For Aim 2, we will recruit a total of 20-40 older adult homebound patients who are likely to be socially isolated, through the Geriatric and General Internal Medicine clinics at Northwestern (over 2,300 homebound older adults) to use the VIPA and accompanying instructional booklet focused on social-isolation. Either the study PI or Research Study Coordinator (RSC) will visit the participant's home, or assist the patient virtually, once consented, to set up the Google Home or Amazon Alexa device for them and review the companion VIPA booklet with them.
  Interventions: Behavioral: VIPA and companion booklet

INTERVENTIONS:
Behavioral: VIPA and companion booklet — Participants will be asked to use the VIPA and accompanying second iteration of the instructional booklet focused on social-isolation. These participants will be surveyed over the phone for 16 weeks (baseline, 2 weeks, 4 weeks, 8 weeks, and 16 weeks) with outcomes measured at each time point.

SUMMARY:
The purpose of this study is to design a companion booklet and pilot test it with a voice-controlled intelligent personal assistants (VIPA), like Google Home or Amazon Alexa, to provide homebound older adult patients with skills and tools to help manage social isolation.

DETAILED DESCRIPTION:
The objective of this pilot study is to design a companion booklet and pilot test it with a voice-controlled intelligent personal assistant (VIPA), Google Home or Amazon Alexa, to provide patients with skills and tools to help manage their social isolation. The companion booklet is a document that will be created using feedback obtained from a panel of geriatric experts, highlighting features of the VIPA that may be most beneficial to socially-isolated older adults. It will be submitted to the IRB for approval once finalized. The specific aims of this project are to:

Aim 1: Design a companion booklet to be used in conjunction with a VIPA (Google Home/Amazon Alexa) for improving social isolation and communication among homebound older adults, defined as someone who is unable to leave the home without assistance of a device or another person, due to a physical or cognitive condition.

Aim 2: Assess the feasibility and implementation of the VIPA (Google Home/Amazon Alexa) and the companion booklet and its impact on clinical and functional outcomes for older adults with social isolation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older;
* Homebound patients of the Northwestern Medicine Geriatrics Program;
* English-speaking; and
* Able to verbally consent

Exclusion Criteria:

* Condition that limits ability to consent, such as severe cognitive impairment or lack of English proficiency
* Less than 65 years of age

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine O'Brien, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VIPA Device and Companion Booklet
Started | 21
Completed (21 participants consented to participate and were enrolled. Two completed their first interviews but were lost to follow up, 3 were unable to connect their devices so were withdrawn, and 1 dropped out after consenting. Therefore, 15 participants completed the study, whereas 17 participants completed the baseline interview and were included in the Overall Number of Baseline Participants section.) | 15
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal due to technical difficulties (see above) | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 17 participants completed the baseline interview, including demographic information, and were included here. However, 2 of those participants were lost to follow up and did not complete the rest of the study. Only 15 participants completed all interviews.
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.53 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Acceptability
Description: usability assessment that we adapted from this original source: Questionnaire for User Interface Satisfaction. Based on: Lund, A.M. (2001) Measuring Usability with the USE Questionnaire. STC Usability SIG Newsletter, 8:2; constructs assessed: usefulness, ease of use, ease of learning, satisfaction. Responses can range from 1 to 7, and scores represent an average of responses so can also range from 1 to 7, with higher scores representing greater acceptability.
Time Frame: 4 weeks, 8 weeks, and 16 weeks
Population: one participant had to miss each of the last two timepoints for logistical reasons
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 15
score on a scale
  4 weeks | 5.2 (1.36)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 5.27 (1.44)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 5.34 (1.53)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.785, ANOVA

2. Primary Outcome: Change in Social Isolation
Description: PROMIS Social Isolation -Short Form 8a: The PROMIS Social Isolation item bank assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others; scores represent T-scores, with a higher score representing higher levels of social isolation. T-score of 50 indicates the population mean, with a standard deviation of 10. In terms of cut points, a T-score of 55-60 represents mild social isolation, 60-70 represents moderate, and >70 represents severe (https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points).
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
T-score
  Baseline | 48.04 (8.54)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 49.44 (8.17)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 47.44 (9.4)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 47.75 (10.93)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.583, ANOVA

3. Primary Outcome: Change in Anxiety
Description: General Anxiety Disorder Scale (GAD-7): Total score (adding all the numbers) provides a possible score from 0-21, higher scores reflect more anxiety.
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
score on a scale
  Baseline | 5.44 (5.85)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 3.87 (4)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 5.57 (4.82)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 3.86 (4.52)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.5015, ANOVA

4. Primary Outcome: Change in Self Efficacy for Managing Social Interactions
Description: PROMIS Self Efficacy for Managing Social Interactions -Short Form 4a: : Confidence in participating in social activities and getting help when necessary. Managing communication with others about their medical condition, including communication with health professionals. Scores represent T-scores, with higher scores representing higher self-efficacy. T-score of 50 indicates the population mean, with a standard deviation of 10. In terms of cut points, a T-score of 30-40 represents low self-efficacy and <30 represents very low (https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points).
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
T-score
  Baseline | 47.59 (8.05)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 48.54 (9.19)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 49.4 (9.18)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 45.96 (8.15)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.3536, ANOVA

5. Primary Outcome: Change in Companionship
Description: PROMIS Companionship -Short Form 4a: The PROMIS adult Companionship item bank assesses perceived availability of someone with whom to share enjoyable social activities such as visiting, talking, celebrations, etc. Scores represent T-scores, with higher scores representing higher levels of companionship. T-score of 50 indicates the population mean, with a standard deviation of 10. In terms of cut points, a T-score of 30-40 represents low companionship and <30 represents very low (https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points).
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
T-score
  Baseline | 48.26 (7.27)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 45.06 (9.03)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 48.72 (7.99)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 46.36 (10.35)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.2688, ANOVA

6. Primary Outcome: Change in Ability to Participate in Social Roles and Activities
Description: PROMIS Ability to Participate in Social Roles and Activities -Short Form 4a: Scores represent T-scores, with higher scores representing a higher perceived ability to participate. T-score of 50 indicates the population mean, with a standard deviation of 10. In terms of cut points, a T-score of 40-45 represents mild difficulty in participating, 30-40 represents moderate, and <30 represents severe (https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points).
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
T-score
  Baseline | 52.97 (6.72)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 50.6 (8.42)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 50.39 (8.23)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 50.04 (7.99)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.728, ANOVA

7. Primary Outcome: Change in Depression
Description: Geriatric Depression Scale (GDS) - Short Form: scores range from 1 to 15, with higher scores reflecting more depressive symptoms.
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
score on a scale
  Baseline | 3.31 (2.65)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 3.8 (3.12)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 2.54 (1.71)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 3.45 (2.7)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.473, ANOVA

8. Primary Outcome: Change in Functional Status
Description: PROMIS-Physical function 8b: PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. Scores represent T-scores, with higher scores representing higher levels of physical function. T-score of 50 indicates the population mean, with a standard deviation of 10. In terms of cut points, a T-score of 40-45 represents mild physical function concerns, 30-40 represents moderate, and <30 represents severe (https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points).
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
T-score
  Baseline | 33.46 (7.82)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 33.18 (6.82)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 31.7 (6.93)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 31.4 (7.99)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.4161, ANOVA

9. Primary Outcome: Change in Cognitive Function
Description: Brief Montreal Cognitive Assessment (MoCA): The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Scores range from 0 to 22, with higher scores representing higher cognitive function. A score of 18 or higher is considered "normal" cognition.
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: after baseline, 1 participant withdrew, and 1 participant missed each of the following timepoints. Only 7 participants completed this measure due to technical difficulties and hearing impairments that impeded participants' ability to complete this measure virtually.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 7
score on a scale
  Baseline | 15.71 (4.31)
  4 weeks: number analyzed (Participants) | 5
  4 weeks | 15 (3.16)
  8 weeks: number analyzed (Participants) | 5
  8 weeks | 16 (4.69)
  16 weeks: number analyzed (Participants) | 5
  16 weeks | 16 (4.04)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.3356, ANOVA

10. Primary Outcome: Change in Well-being
Description: Neuro-QOL Positive Affect & Well-Being: Scores represent T-scores, and higher scores indicate better self-reported well-being. T-score of 50 indicates the population mean, with a standard deviation of 10. In terms of cut points, a T-score of 30-40 represents low positive affect and <30 represents very low (https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/promis-score-cut-points).
Time Frame: baseline, 4 weeks, 8 weeks, and 16 weeks
Population: one participant withdrew after baseline, and one participant missed each of the final two timepoints
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | VIPA Device and Companion Booklet
Number analyzed (Participants) | 16
T-score
  Baseline | 54.27 (7.25)
  4 weeks: number analyzed (Participants) | 15
  4 weeks | 54.73 (7.08)
  8 weeks: number analyzed (Participants) | 14
  8 weeks | 55.21 (9.32)
  16 weeks: number analyzed (Participants) | 14
  16 weeks | 54.66 (9)
Statistical Analysis 1: Comparison: VIPA Device and Companion Booklet; Test type: Other; p = 0.9825, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | VIPA Device and Companion Booklet
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT04900272/Prot_000.pdf
  • Informed Consent Form (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT04900272/ICF_001.pdf